CLINICAL TRIAL: NCT06511778
Title: sTErnAl heMostasiS Trial (TEAMS Trial)
Brief Title: sTErnAl heMostasiS Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: WakeMed Health and Hospitals (Other)
Collaborators: Dilon Technologies (Unknown)
Responsible Party: Principal Investigator, Judson Williams, Principal Investigator, WakeMed Health and Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TEAMS
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Excessive Bleeding During Surgery

STUDY DESIGN:
Intervention Model Description: Patients undergoing on pump sternotomy surgery
Who Masked: Participant
Masking Description: The patient will not know whether they had the hemostatic agent applied during scheduled on pump sternotomy surgery as an additional adjunct to control bleeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Application of Hemoblast Hemostatic Agent (No Intervention): Patients who are randomized to "control" will not receive application of the Hemoblast hemostatic agent during on pump sternotomy surgery.
- Application of Hemoblast Hemostatic Agent (Active Comparator): Patients who are randomized to "treatment" will receive application of the Hemoblast hemostatic agent during on pump sternotomy surgery.
  Interventions: Drug: Hemoblast Bellows application

INTERVENTIONS:
Drug: Hemoblast Bellows application — Hemoblast bellows is a hemostatic agent clinically proven effective on the validated SPOT GRADE scale for minimal, mild, and moderate bleeding. Patients will have the Hemoblast bellows applied during on pump sternotomy surgery.
  Arms: Application of Hemoblast Hemostatic Agent

SUMMARY:
Sternal bleeding remains an unsolved problem for cardiac surgery teams costing operative time, blood loss, and distraction from the critical operative field. As such, the following is an investigator-initiated trial to determine whether application of a topical hemostatic agent reduces sternal bleeding during cardiac surgery using sternotomy approach.

DETAILED DESCRIPTION:
This is a prospective randomized 1:1 trial to evaluate the efficacy of the application of HEMOBLASTTM during cardiothoracic surgery to reduce the increased risk of sternal bleeding in 30 treatment and 30 control patients.

Enrollment will be open to all eligible participants undergoing cardiothoracic surgery who sign an informed consent.

The study will also collect demographic data and relevant clinical data, such as medical history, diagnosis, family history, laboratory data, radiological images and reports, and diagnostic procedure reports.

All enrolled subjects will be followed during their hospitalization until discharge for bleeding complications after their surgical procedure as well as a sternal bleeding SPOT GRADE TM score will be recorded independently by both the cardiac surgeon and assisting cardiothoracic PA-C, before and after the application of the topical hemostatic agent. There will be no restriction on the use of electrocautery or vancomycin paste as existing routine adjuncts used in cardiothoracic surgery for sternal hemostasis. Chest tube output measurements will be collected at 6, 12, and 24 hours postoperatively. The patients will be assessed at the time of hospital discharge for any complications related to sternal or intrathoracic bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients are scheduled to undergo on-pump open chest cardiothoracic surgery.
* Patients must be willing and able to provide written informed consent.
* If the patient is of childbearing potential, they must have a negative pregnancy test within 24 hours of the index procedure.
* Patients must be at least 21 years of age.
* Patients have at least one of the following risk factors:

  1. Undergoing redo sternotomy
  2. Have a preoperative platelet count <150 mg/dL
  3. Are on dual antiplatelet therapy (blood thinners) < 5 days prior to sternotomy
  4. Have a BMI (body mass index)> 35
  5. Are undergoing combined CABG (coronary artery bypass surgery)/valve surgery
  6. Have chronic kidney disease (GFR <60 ml/min) or ESRD (end stage renal disease)

Exclusion Criteria:

* Patients who undergo thoracotomy approach
* Patients who are not deemed an appropriate candidate by the investigator.
* Patients who are pregnant or nursing, or who plan to become pregnant during the course of this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sternal Bleeding Score | Sternotomy creation
  A sternal bleeding score will be performed independently by surgeon and physician assistant utilizing the SPOT GRADE bleeding scale ranging from 0-5. 0 (no bleeding), 1 (minimal bleeding), 2 (mild bleeding), 3 (moderate bleeding), 4 (severe bleeding), 5 (extreme bleeding) before and after hemostatic agent application
Sternal Bleeding Score | Sternal closure
  A sternal bleeding score will be performed independently by surgeon and physician assistant utilizing the SPOT GRADE bleeding scale ranging from 0-5. 0 (no bleeding), 1 (minimal bleeding), 2 (mild bleeding), 3 (moderate bleeding), 4 (severe bleeding), 5 (extreme bleeding)
Reoperation for Bleeding | Through hospitalization, average of 6 days
  Patients will be monitored for incidences of reoperation due to bleeding
Chest Tube Output | 6 hours postoperatively
  The patient's chest tube output will be recorded after surgery

SECONDARY OUTCOMES:
Chest Tube Output | 12 and 24 hours postoperatively
  The patient's chest tube output will be recorded after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- WakeMed Health and Hospitals, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HEMOBLAST™ Bellows Hemostatic Agent [instructions for use]. Dilon Technologies, Inc.
- [Background] Spotnitz WD, Zielske D, Centis V, Hoffman R, Gillen DL, Wittmann C, Guyot V, Campos DM, Forest P, Pearson A, McAfee PC. The SPOT GRADE: A New Method for Reproducibly Quantifying Surgical Wound Bleeding. Spine (Phila Pa 1976). 2018 Jun 1;43(11):E664-E671. doi: 10.1097/BRS.0000000000002447. PMID 29019803
- [Background] Now That's Real Stopping Powder [Information Brochure]. Dilon Technologies, Inc.
- [Background] Elassal AA, Al-Ebrahim KE, Debis RS, Ragab ES, Faden MS, Fatani MA, Allam AR, Abdulla AH, Bukhary AM, Noaman NA, Eldib OS. Re-exploration for bleeding after cardiac surgery: revaluation of urgency and factors promoting low rate. J Cardiothorac Surg. 2021 Jun 7;16(1):166. doi: 10.1186/s13019-021-01545-4. PMID 34099003